CLINICAL TRIAL: NCT00823329
Title: Calorie Balance Monitoring and Analysis of Body Composition and Hydration
Brief Title: Calorie Balance Monitoring and Analysis of Body Composition and Hydration Status
Acronym: PCMMS
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Ori Diagnostic Instruments LLC (Other)
Responsible Party: Zsolt Ori, MD, MS, FACP, Ori Diagnostic Instruments L.L.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ORI-DGI-001
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Energy Metabolism; Energy Expenditure; Body Composition; Body Fluids
Keywords: measurement of energy expenditure of physical activity; analysis of body composition and hydration status
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: cardiac stress testing with an exercise machine — Standardized graded cardiac stress testing with an exercise machine will be performed according to the protocol of the American Heart Association

SUMMARY:
The investigators are developing two new medical instruments: 1. the Intelligent Sensor Belt (ISB), and 2. the Body Composition and Hydration Status Analyzer (BC-HS-A). ISB serves the purpose of measuring calorie/ energy consumption of the human body during physical activity. The BC-HS-A measures the body composition, i.e. the fat and lean body mass and the hydration status i.e the amount of water inside and outside of the body cells.

The goal of this pilot study is to obtain data from the investigators prototype medical instruments: 1. ISB, and 2. BC-HS-A during physical exercise and compare those results with readings of other commercially available instruments or exercise equipments. The investigators would be testing for technical feasibility and, through comparison with existing measuring devices, the reliability of the investigators prototype.

DETAILED DESCRIPTION:
Our goal is the development of a non-invasive, Portable Comprehensive Metabolic Monitoring System (PCMMS) for continuous measurement and monitoring of parameters of the human energy metabolism.

The current project focuses on the development of two hardware components of PCMMS: 1. the Intelligent Sensor Belt (ISB), and 2. the Body Composition (BC) & Hydration Status (HS) Analyzer (BC--HS-A).

ISB is designed to be worn around the chest or waist and measures the energy expenditure of physical activity (PAE) via sensors for heart rate, tri-axial acceleration, and temperature.

BC-HS-A utilizes multi-frequency bio-impedance measurements through electrodes attached to one hand and opposite foot. This instrument is not used continuously but intermittently when momentary values of BC and HS are desired.

This pilot study is designed to obtain data from our instruments during a limited exercise session to gage its function and to determine its feasibility for the intended use. The pilot study will be performed on healthy volunteers who would wear ISB during a graded cardiac stress testing on various exercise machines such as the stationary bicycle, treadmill, stair case, and rowing machine. PAE measured by ISB will be compared with the estimated results of the particular exercise equipment. The BC measuring function of our BC-HS-A will be compared with a commercially available bioimpedance analyzer. Changes of hydration status during exercise measured by our BC-HS-A will be compared against precision measurements of body weight before and after exercise estimating total water loss of the body. All results will be reported in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* interested participants who have maintained the same weight for several months and are healthy, are not pregnant and not wanting to become pregnant during the study period, do not take any drugs, and exercise regularly to maintain their weight will be invited.

Exclusion Criteria:

* patients taking medication for bodily illness/disease, women who are pregnant or wanting to become pregnant during the study period, and those who have not followed a regular exercise regimen will not be included in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-10; Primary Completion 2012-10; Study Completion 2012-10

PRIMARY OUTCOMES:
Comparison of the measuring function of our prototype devices with that one of commercially available measuring instruments | The outcome is assessed within few weeks of actual testing

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt P Ori, MD, Principal Investigator — Boone Hospital Center
Locations (1):
- McKee Gym of the Department of Nutrition and Exercise Physiology, Columbia, Missouri, United States